CLINICAL TRIAL: NCT06158581
Title: The Emotion Awareness and Skills Enhancement (EASE) Program Versus the Unified Protocol (UP)
Brief Title: Comparing Two Different Emotion Therapies for Autistic Youth and Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Alabama, Tuscaloosa (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Carla Mazefsky, Professor of Psychiatry, Psychology, and Clinical and Translational Science, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY23090024; IDD-2022C1-26418 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A rater blind to condition assignment will assign CGI ratings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Emotion Awareness and Skills Enhancement (Experimental): EASE is a 16-session mindfulness-based intervention (MBI). It emphasizes a small set of core concepts (i.e., mindfulness practices, distress tolerance, encouraging helpful thoughts, self-compassion) that are repeated with consistent language throughout. Emphasis is placed on increasing awareness of gradients of emotional arousal.
  Interventions: Behavioral: The Emotion Awareness and Skills Enhancement Program
- The Unified Protocol (Active Comparator): UP is a 12-21 session cognitive behavioral therapy (CBT) based treatment. In this study, there will be 16 sessions. UP is focused on identifying emotions and building new coping strategies. It is customizable to meet the needs of the individual.
  Interventions: Behavioral: The Unified Protocol

INTERVENTIONS:
Behavioral: The Emotion Awareness and Skills Enhancement Program — EASE is a cutting-edge program created by researchers at the University of Alabama and the University of Pittsburgh in collaboration with autistic individuals, caregivers of autistic youth, and therapists. The overarching goal of the program is to support autistic clients who want to work on emotion regulation. EASE is unique because it targets emotional distress in autistic youth and adults, instead of targeting the core symptoms of autism (i.e., it is not a social skills intervention).
  The program is a 16-session, mindfulness-based intervention. Each session is 1:1 for 45 minutes to one hour. While the program is designed for individual intervention, caregivers are also invited to play an active role on the care team.
  Other Names: EASE
  Arms: The Emotion Awareness and Skills Enhancement
Behavioral: The Unified Protocol — UP is a thoroughly-studied, manualized intervention created by researchers at the University of Miami in conjunction with researchers at Boston University. The program was designed to be customizable to meet the needs of people with a variety of diagnoses, allowing more individuals to access emotion regulation resources. The protocol also has different modules to accommodate different developmental levels (UP-Children, UP-Adolescent, UP-Adult). The overall goal of UP is to help clients identify emotions and build new strategies to cope with stressful life situations and distressing emotions.
  The protocol is flexible, with each session is about 45 to 60 minutes and the number of sessions varying between 12 - 21 sessions. For the current study, the treatment will take place over 16 sessions. The intervention is cognitive behavioral therapy (CBT) based but also includes hints of mindfulness-based intervention strategies.
  Other Names: UP
  Arms: The Unified Protocol

SUMMARY:
Too few clinicians are able and willing to help autistic patients. A recent review identified challenges to mental health service delivery in autism, including a lack of interventions designed for community implementation and limited workforce capacity. It has been argued that improving impairment in emotion regulation has the potential to improve a range of mental health difficulties in autistic people. In this clinical trial, the investigators are comparing two evidence-based interventions for emotion regulation, to determine if one created specifically for autistic people is clinically superior. The interventions will be implemented in the community, through partnering agencies.

DETAILED DESCRIPTION:
This study will compare the effectiveness of two transdiagnostic interventions for autistic adolescents and young adults - an intervention in widespread use among non-autistic populations (The Unified Protocol; UP) versus an autism-specific intervention (The Emotion Awareness and Skills Enhancement Program; EASE). The UP and EASE are ideal comparators because they are structurally equivalent and transdiagnostic - both shown to improve mental health outcomes that stakeholders identify as important, such as depression, irritability, and anxiety. The investigators will partner with 10 different community clinics in Pennsylvania and Alabama to recruit participants and facilitate the interventions. Each clinic will be randomized to use either UP or EASE. The investigators will look at effectiveness of the treatments, as well as the feasibility, benefits and harms.

ELIGIBILITY:
Inclusion Criteria:

* professional diagnosis of ASD
* a score in the clinical range on the EDI-Reactivity or EDI-Dysphoria scale based on caregiver report or self-report
* The study is open to people with a range of communication abilities. Participants must be able to consent to the study themselves and answer questions about themselves.
* Participants need to have a support person that could answer questions about them too. This could be a parent, caregiver, family member, partner or friend.
* Participants must live in Alabama or Pennsylvania.

Exclusion Criteria:

- Higher level of care is needed (Imminent Suicide / Homicide Threat, acute psychosis, mania)

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 470 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Emotion Dysregulation Inventory | Baseline, Midpoint (after completing 8 sessions), Post treatment (after all 16 sessions, average 16-20 weeks), 3 months following post-treatment
  The EDI does not have a single overall score. It is comprised of two scales: Reactivity and Dysphoria. Items are on a 0 to 4 scale, where 0 is Never happens and 4 is Almost always happens or causes a serious problem. There are clinical cutoffs for both scales.
Weiner's Acceptability, Appropriateness, & Feasibility of Intervention Scales | Baseline and Post treatment of first client (after all 16 sessions, average 16-20 weeks)
  Weiner's is a widely used 12-item battery of three scales assessing intervention acceptability, appropriateness, and feasibility with strong psychometric properties. There is a 1 to 5 scale, where 1 is Completely disagree and 5 is Completely agree. Higher scores indicate greater acceptability, appropriateness, and feasibility.
Provider Self-Efficacy Scale | Baseline and Post trial (4 years)
  It assesses both knowledge (of protocol) and confidence (in one's ability to implement as intended). It is a 0-10 scale, where 0 is not at all confident and 10 is extremely confident. Higher scores indicate higher confidence.

SECONDARY OUTCOMES:
Clinical Global Impressions | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks)
  The CGI will be used as a measure of overall improvement. The CGI was designed to measure overall symptomatic change at a specific time as compared to baseline that is completed by a rater who is blind to treatment assignment. Scores range from 1 (Very Much Improved) to 4 (Unchanged) to 7 (Very Much Worse). It is only a single item, and lower scores indicate more improvement.
PROMIS Depression | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks), 3 months following post-treatment
  It is a brief, change sensitive 8 item measure. It is a 1-5 scale, where 1 is Never and 5 is Always.
PROMIS Anxiety | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks), 3 months following post-treatment
  It is a brief, change sensitive 8 item measure. It is a 1-5 scale, where 1 is Never and 5 is Always.
Buss-Perry Aggression Questionnaire | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks), 3 months following post-treatment
  27-item self-report measure of general aggression, physical aggression, verbal aggression, anger, and hostility. It is a 1-7 scale, where 1 is Extremely uncharacteristic of me and 7 is Extremely characteristic of me.
Emotion Regulation Questionnaire for Children and Adolescents | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks), 3 months following post-treatment
  ERQ-CA has10 items that comprise of two scales: cognitive reappraisal use and expressive suppression, which are two regulatory strategies considered adaptive and protective in terms of mental health. It is a 1-7 scale, where 1 is Strongly disagree and 7 is Strongly agree.
Child & Adolescent Mindfulness Measure | Baseline, Midpoint (after completing 8 sessions), Post treatment (after all 16 sessions, average 16-20 weeks)
  CAMM is a 10-item self-report measure of mindfulness. It is a 0-4 scale, where 0 is Never true and 4 is Always true. When scoring, you reverse all scores (i.e. 0 to 4) and then sum. Higher scores correspond to higher levels of mindfulness.
WHO Quality of Life-BREF-ID | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks), 3 months following post-treatment
  WHOQoL-BREF-ID is a simplified version of the World Health Organization Quality of Life. It has a 3 or 5 point visual response scale, where 1 is Not at all and 5 is Totally.
Satisfaction with Life Scale | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks)
  Satisfaction was Life Scale is a 5-item measure of global life satisfaction. It is a 1-7 scale, where 1 is Strongly disagree and 7 is Strongly agree.
Self-Compassion Scale-Youth Version | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks), 3 months following post-treatment
  Self-Compassion Scale - Youth Version consists of 17 self-report items ranked on a 5-point Likert scale, yielding six subscales (self-kindness, self-judgment, common humanity, isolation, mindfulness, over-identification) and an overall score. 1 is Almost Never and 5 Almost Always.
Relationships, Employment, Autonomy, and Life Satisfaction | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks)
  REALS Measures are a compilation of scales tapping many areas of adult life. Each scale is scored independently and should be utilized as different sources of information. It does not produce a global outcome score. With the frequency scales, it is a 0-4 scale where 0 is Never and 4 is Always.
AASPIRE Flourishing Scale | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks), 3 months following post-treatment
  It is 9 item scale that assesses aspects of life satisfaction for autistic individuals. It is a scale from strongly disagree to strongly agree.
AASPIRE Burnout Scale Short Form | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks), 3 months following post-treatment
  It is a 14-item self-report measure of autistic burnout. It is a scale from strongly disagree to strongly agree.
Credibility and Expectancy Questionnaire | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks)
  It will assess treatment expectancy and rationale for the assessed treatments.
AASPIRE Patient Health Questionnaire-9 | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks), 3 months following post-treatment
  This is a 9-item self-report questionnaire for screening, diagnosing, monitoring and measuring the severity of depression, that includes an item that is widely utilized as an index of suicidal ideation severity. Each item is rated on a scale from Rarely or not at all to Almost every day. Higher scores would relate to higher depression.
Inventory of Statements about Self-Injury | Baseline, Post treatment (after all 16 sessions, average 16-20 weeks), 3 months following post-treatment
  ISAS is a continuous self-report measure of self-injurious behaviors. It is the most commonly used measure of self-injury. Higher numbers in Section 1 would indicate more self-injurious behaviors.
Working Alliance Inventory | Midpoint (after completing 8 sessions, average 8 weeks), After completing 15 sessions (average 15-19 weeks)
  WAI is a clinician-report measure assessing the therapeutic alliance between the client/participant and the clinician. The measure is 12 items, rated on a 5-point scale.
Vanderbilt Therapeutic Alliance Scales Revised, Short Form | 2 randomized timepoints over up to 20 Weeks
  VTAS-R-SF is an observational measure of alliance and consists of five items to capture the strength of the perceived support and trust, participation, and agreement on tasks and goals between client and therapist. Each item is rated 0-5, and higher scores mean more alliance. The measure is used for coding videos of the therapy sessions. It will be completed twice with each participant but the timepoint is randomized (one randomized session from the first half of therapy and one randomized session from the second half of therapy).
Child Involvement Rating Scale | 2 randomized timepoints over up to 20 Weeks
  Child Involvement Rating Scale is a 10-item, 6-point observational scale to rate involvement and engagement during therapy. The first 6 items rate positive involvement where 0 is not at all and 5 is a great deal. The last 4 items rate negative involvement where 0 is not at all and 5 is a great deal. The measure is used for coding videos of the therapy sessions. The measure will be completed twice with each participant but the timepoint is randomized (one randomized session from the first half of therapy and one randomized session from the second half of therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Carla Mazefsky, PhD, Principal Investigator — University of Pittsburgh; Susan White, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama, Tuscaloosa, Alabama
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
PCORI, the funder, is committed to open science and the investigators are required to deposit their Full Data package in a PCORI-designated data repository. The investigators will enter into a Data Contributor Agreement with a PCORI-designated repository after the investigators complete data collection. The repository will make the Full Data Package available for third-party requests when PCORI makes the Final Research Report available on the PCORI website, or at the time of publication of the research project's primary results in a peer-reviewed journal, whichever comes first.
Time Frame: The data will be uploaded to the repository by December 2027.
Access Criteria: Investigators must submit a data request to the PCORI-designated repository. If the request is approved, the data requestor's institution must enter into a Data Use Agreement with the repository. If the investigators receive requests for data directly from a third party, the investigators will need to notify PCORI if the data is not yet in the repository.

REFERENCES:
- [Background] Conner CM, White SW, Beck KB, Golt J, Smith IC, Mazefsky CA. Improving emotion regulation ability in autism: The Emotional Awareness and Skills Enhancement (EASE) program. Autism. 2019 Jul;23(5):1273-1287. doi: 10.1177/1362361318810709. Epub 2018 Nov 7. PMID 30400749
- [Background] Ellard KK, Fairholme CP, Boisseau CL, Farchione TJ, Barlow DH. Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders: Protocol Development and Initial Outcome Data. Cogn Behav Pract. 2010 Feb;17(1):88-101. doi: 10.1016/j.cbpra.2009.06.002. Epub 2010 Jan 29. PMID 33762811
- [Background] Barlow DH, Farchione T, Sauer-Zavala, Shannon Murray Latin H, et al. Unified Protocol for Transdiagnostic Treatment of Emotional Disorders: Therapist Guide. Second Edi. Oxford University Press; 2017.
- [Background] Ehrenreich-May J, Kennedy SM, Sherman JA, et al. Unified Protocols for Transdiagnostic Treatment of Emotional Disorders in Children and Adolescents: Therapist Guide. Oxford University Press; 2017.